CLINICAL TRIAL: NCT03447145
Title: Phase I Study of Tolerance and Pharmacokinetics of TQ-B3203
Brief Title: A New Drug Used for Advanced Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3203-I-01
Record Dates: First submitted 2017-12-26; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3203 (Experimental)
  Interventions: Drug: TQ-B3203

INTERVENTIONS:
Drug: TQ-B3203 — dose escalation, 2/4/6/10/14/18mg/m2

SUMMARY:
To identify the safety and tolerance of TQ-B3203.

ELIGIBILITY:
Inclusion Criteria:

* Patients definitedly diagnosed by pathology and/or cytology as advanced solid tumor,those who lack of standard treatments or treatment failure;
* Patients treated with chemotherapy agents or surgery before being enrolled into the study need waiting for 30 days, 6 weeks will be needed if agents were Nitrocarbamide and Mitomycin C
* 18-70 years old,Eastern Cooperative Oncology Group(ECOG):0-1,Life expectancy of more than 3 months,BMI:18.5-26;
* Main organs function is normal;
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped;
* Patients should be voluntary and sign the informed consents before taking part in the study;

Exclusion Criteria:

* Patients with Malignant tumors within 5 years, except for non-melanoma skin cancer and in situ cancer;
* Patients who participated in other anticancer drug clinical trials within 4 weeks;
* Patients treated with Irinotecan,Topotecan and any other topoisomerase I inhibitors or related clinical trials;
* Patients of double locus mutation of UGT1A1*6、UGT1A1*28;
* Patients who cannot stop using inhibitors of CYP3A4 and UGT1A1 7 days before enrolled in the study,inducers of CYP3A4 need 2 weeks.
* Patients who can not be injected and patients with interstitial pneumonia or radiation pneumonia;
* Patients with pericardial effusion,pleural effusion or ascitic fluid, patients with 2nd respiratory syndrome or above are refused according to National Cancer Institute Common Terminology Criteria for Adverse Events(CTC AE);
* Patients with brain metastasis, spinal cord compression, cancerous meningitis, CT or MRI examination reminds patients with cerebral or soft meningeal diseases in the screening phase;
* Patients with drug abuse history or unable to get rid of drugs or Patients with mental disorders;
* Patients with non-healing wounds or fractures;
* Patients got radiotherapy for bone metastases 2 weeks before being enrolled in the study;
* Patients with urine pro 2+ and the quantitative result>1.0g
* Patients got Arteriovenous thrombosis 6 months before being the study "Blood pressure unable to be controlled ideally by one drug(systolic pressure≥150 mmHg，diastolic pressure≥90 mmHg);
* Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias or cardiac insufficiency (including QTc≥480ms) and patients with Grade 3 or higher congestive heart failure (NYHA Classification);"
* Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history;
* Patients with thyroid dysfunction;
* Patients diagnosed with glaucoma,or prostatomegaly need to be treated;
* Coagulation function abnormality: haemorrhagic tendencies (e.g. active digestive tract ulcer), or are receiving thrombolytic or anticoagulant therapy
* Patients with concomitant diseases which could seriously endanger themselves or those who won't complete the study according to investigators;
* Patient with hepatitis b surface antigen positive(HBV DNA>1000) or hepatitis C virus(HCV);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-12-26 (Estimated); Study Completion 2018-12-26 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose(MTD) | 21 days
dose-limiting toxicity(DLT) | 21 days
Peak Plasma Concentration(Cmax) | 21 days
Peak time（Tmax） | 21 days
Half life（t1/2） | 21 days
Area under the plasma concentration versus time curve (AUC) | 21 days
Clearance（CL） | 21 days

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | each 42 days up to intolerance the toxicity or progression disease (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China